CLINICAL TRIAL: NCT03890705
Title: Postpartum Family Planning Utilization and Associated Factors Among Women During the First Year After Childbirth in Assiut District
Brief Title: Postpartum Family Planning Utilization and Associated Factors Among Women During First Year After Childbirth in Assiut
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maria Adel Zaky, principal investigator, Assiut University
Other Study IDs: Family planning Assiut
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- postpartum women: Women aged (15-49) and had given birth in the past 12 months

SUMMARY:
Postpartum family planning is defined as prevention of unintended pregnancy and closely spaced pregnancies during the first 12 months after the child birth postpartum contraceptive utilization is important because some women resume ovulation after 28 days postpartum inter-pregnancy intervals shorter than 18 to 24 months have been associated with an increased risk of fetal and maternal deaths ,35% of children younger than five deaths could be avoided if births spaced 36 months

DETAILED DESCRIPTION:
According to Egyptian demographic health survey , unmet need for family planning increased from 11.6% in 2008 to be 12.6% in 2014, contraception prevalence rate decreased from 60% in 2008 to 59% in 2014.

In Assiut Contraception prevalence rate decreased form 47.4 in 2008 to 41.4 in 2014 Total fertility rate increased from 3 in 2008 to 3.5 children/woman in 2014, Assiut Total fertility rate was 4.2 children/woman in 2014 . projections for the year 2030 estimated that total fertility rate would decline to be 2.1 births/woman if Contraceptive prevalence rate could rise to be 74.4% .

Routine childhood immunization services include more than 500 million regular contacts annually, most women seek child immunization for their children so each immunization represents an opportunity to reach women with Postpartum family planning counselling so World Health Organization recommends Postpartum family planning as a critical healthcare component and World Contraception Day 26 September 2018, Met the theme"Postpartum family planning: essential for ensuring woman health and their babies" World Health Organization for family planning research agenda listed postpartum family planning utilization as a higher priority score with score 83.90

ELIGIBILITY:
Inclusion Criteria:

* Women aged (15-49)
* and had given birth during the past 12 months.

Exclusion Criteria:

* Women that had children older than 12 months
* Pregnant women
* Sexually inactive women as widow and divorced
* Women who had done abdominal hysterectomy

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Women aged (15-49) who had given birth during the past 12 months
Study Population: Women aged (15-49) who had given birth during the past 12 months and attending the Primary health care units for child immunization at the age of 12 months
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
postpartum family planning utilization rate questionnaire | one year
  postpartum contraceptive utilization rate among women during first year postpartum in Assiut district

SECONDARY OUTCOMES:
factors affecting postpartum family planning utilization questionnaire | one year
  factors affecting postpartum family planning utilization among women who had given birth during the past 12 months in Assiut district

CONTACTS AND LOCATIONS:
Overall Officials: maria tadros, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Jackson E, Glasier A. Return of ovulation and menses in postpartum nonlactating women: a systematic review. Obstet Gynecol. 2011 Mar;117(3):657-662. doi: 10.1097/AOG.0b013e31820ce18c. PMID 21343770
- [Background] Ministry of Health and Population [Egypt], El-Zanaty and Associates [Egypt], and ICF International. 2015. Egypt Demographic and Health Survey 2014. Cairo, Egypt and Rockville, Maryland, USA: Ministry of Health and Population and ICF International.
- [Background] El-Masry R et al. Unmet need for family planning among women in rural Egypt International Journal of Community Medicine and Public Health. 2018 Apr;5(4):1252-1261
- [Background] Ali M, Seuc A, Rahimi A, Festin M, Temmerman M. A global research agenda for family planning: results of an exercise for setting research priorities. Bull World Health Organ. 2014 Feb 1;92(2):93-8. doi: 10.2471/BLT.13.122242. Epub 2013 Nov 4. PMID 24623902
- See also: integration of family planning with immunization services by united states agency international development — https://www.fhi360.org/sites/default/files/media/documents/integration-family-planning-immunization.pdf
- See also: Programming strategies for Postpartum Family Planning — https://apps.who.int/iris/bitstream/handle/10665/93680/9789241506496_eng.pdf?sequence=1